CLINICAL TRIAL: NCT01453166
Title: The Effect of Brazilian Heart Prevent Meal Program Accessible for the Population to Prevent New Cardiovascular Events: A Pilot Randomized Clinical Trial
Brief Title: Brazilian Heart-Prevent Meal - A Pilot Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital do Coracao (Other)
Collaborators: Ministry of Health, Brazil (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 01/2011
Record Dates: First submitted 2011-10-11; First posted 2011-10-17 (Estimated); Results first posted 2012-07-17 (Estimated); Last update posted 2012-07-19 (Estimated); Status verified 2012-07

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 (Experimental): Nutrient profile of the diets used was based on the Brazilian guidelines to cardiovascular disease treatment.The main difference between this group involves a Brazilian version of accessible and energy density concept dietary therapy to cardiovascular diseases. Furthermore, it explores a set of tools and educational materials that help the patient understand and follow the principles of balanced and healthy diet weekly session with the dietitians which could be in person, by phone or in a gourmet shop. During attendances at the gourmet shop, patients received tips for eating in restaurants, instruction on label reading and a list of typical foods. The menus were based on typical foods consumed in Brazil, all foods included in the menu were low-cost and widely available at local markets
  Interventions: Other: Brazilian heart-prevent meal
- Group 2 (Experimental): Group B received the usual dietary therapy to patients with cardiovascular diseases, which had the same nutrient profile as presented in Group A, but customized by the integration of mediterranean typical foods (e.g. olive oil and nuts). The difference between groups B and C was the number of sessions with the dietician. Group B received weekly sessions, which could be in person or by phone, and group C had monthly in person sessions
  Interventions: Other: Heart prevent control meal weekly
- Group 3 (Experimental): Group C received the usual dietary therapy to patients with cardiovascular diseases, which had the same nutrient profile as presented in Group A and B, but customized by the integration of mediterranean typical foods (e.g. olive oil and nuts) at the same of group B. The difference of group C was the number of sessions with the dietician. That happen monthly in person sessions.
  Interventions: Other: Heart prevent control Meal monthly

INTERVENTIONS:
Other: Brazilian heart-prevent meal — Nutrient profile of the diets used was based on the Brazilian guidelines to cardiovascular disease treatment.The main difference between this group involves a Brazilian version of accessible and energy density concept dietary therapy to cardiovascular diseases. Furthermore, it explores a set of tools and educational materials that help the patient understand and follow the principles of balanced and healthy diet weekly session with the dietitians which could be in person, by phone or in a gourmet shop. During attendances at the gourmet shop, patients received tips for eating in restaurants, instruction on label reading and a list of typical foods. The menus were based on typical foods consumed in Brazil, all foods included in the menu were low-cost and widely available at local markets
  Other Names: Dietetic intervation developed by reseachers
  Arms: Group 1
Other: Heart prevent control meal weekly — received the usual dietary therapy to patients with cardiovascular diseases, which had the same nutrient profile as presented in Group A, but customized by the integration of mediterranean typical foods (e.g. olive oil and nuts). The difference between groups B and C was the number of sessions with the dietician. Group B received weekly sessions, which could be in person or by phone, and group C had monthly in person sessions
  Other Names: Dietetic intervation
  Arms: Group 2
Other: Heart prevent control Meal monthly — received the usual dietary therapy to patients with cardiovascular diseases, which had the same nutrient profile as presented in Group A and B, but customized by the integration of mediterranean typical foods (e.g. olive oil and nuts) at the same of group B. The difference of group C was the number of sessions with the dietician. That happen monthly in person sessions.
  Other Names: Dietetic intervation once per month
  Arms: Group 3

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a brazilian cardioprotective diet plan to reduce cardiovascular risk factors of new cardiovascular events.

DETAILED DESCRIPTION:
Cardiovascular diseases are the leading cause of mortality in both sexes in Brazil and worldwide. Modifying risk factors such as diet and lifestyle can prevent most cases of cardiovascular disease. This pilot trial is based on specific and traditional brazilian food. The objective is to reduce risk factors such as obesity, high blood pressure,dyslipidemia and diabetes in patients with cardiovascular disease history.

ELIGIBILITY:
Inclusion Criteria:

* Any coronary artery disease evidence in the past 10 years; or any ischemic stroke or TIA evidence in the past 10 years; or peripheral arterial disease in the past 10 years; or at least one of the following additional risk factors:
* Diabetes Mellitus; Hypertension; Dyslipidemia; Coronary artery disease family history;
* Asymptomatic carotid artery disease;
* Body mass index> 25 kg/m2 for adults and> 28 kg/m2 for seniors

Exclusion Criteria:

* Neurocognitive or psychiatric condition;
* Life expectancy less than 6 months (eg, metastatic malignancy or other defined as clinical trial investigators).
* Pregnancy or breast feeding.
* Hepatic impairment defined as elevated liver enzymes above three times the upper limit of normal
* Renal impairment defined as creatinine values higher than 1.5 mg/dL.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2011-09; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernardete Weber, PhD, Principal Investigator — Hospital do Coração
Locations (1):
- Hospital do Coracao, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Weber B, Galante AP, Bersch-Ferreira AC, Torreglosa CR, Carvalho VO, Victor Eda S, Espirito-Santo JA, Ross-Fernandes MB, Soares RM, Costa RP, Lara Ede S, Buehler AM, Berwanger O. Effects of Brazilian Cardioprotective Diet Program on risk factors in patients with coronary heart disease: a Brazilian Cardioprotective Diet randomized pilot trial. Clinics (Sao Paulo). 2012 Dec;67(12):1407-14. doi: 10.6061/clinics/2012(12)10. PMID 23295594

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 151 patients agreed to participate of the screening day in the Hospital do Coração in São Paulo Brazil. After eligibility set, From September 2011 to December 2011,122 patients were randomized for one of three treatment groups
Pre-assignment Details: Of those ineligible, 9 missed the screening day, 14 did not present previews cardiovascular event, 3 declined to participate. After randomization, two patients were identified as ineligible to present chronic renal and hepatic insufficiency, and three dropped out of the study Among those who met inclusion criteria, 117 participants completed study
Groups:
- Brazilian Heart-prevent Meal: Nutrient profile of the diets used in the three groups was based on the Brazilian guidelines to cardiovascular disease treatment.The main difference between this group involves a Brazilian version of accessible and energy density concept dietary therapy to cardiovascular diseases. Furthermore, it explores a set of tools and educational materials that help the patient understand and follow the principles of balanced and healthy diet weekly session with the dietitians which could be in person, by phone or in a gourmet shop. During attendances at the gourmet shop, patients received tips for eating in restaurants, instruction on label reading and a list of typical foods. The menus were based on typical foods consumed in Brazil, prioritizing the Brazilian culture and regional habits. All foods included in the menu were low-cost and widely available at local markets
- Heart Prevent Meal I: Group B received the usual dietary therapy to patients with cardiovascular diseases, which had the same nutrient profile as presented in Group A, but customized by the integration of mediterranean typical foods (e.g. olive oil and nuts). The difference between groups B and C was the number of sessions with the dietician. Group B received weekly sessions, which could be in person or by phone, and group C had monthly in person sessions
- Heart Prevent Meal II: Group C received the usual dietary therapy to patients with cardiovascular diseases, which had the same nutrient profile as presented in Group A and B, but customized by the integration of mediterranean typical foods (e.g. olive oil and nuts) at the same of group B. The difference of group C was the number of sessions with the dietician. That happen monthly in person sessions.
Period: Overall Study
Arm/Group | Brazilian Heart-prevent Meal | Heart Prevent Meal I | Heart Prevent Meal II
Started | 42 | 41 | 39
Completed | 40 | 39 | 38
Not Completed | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Brazilian Heart-prevent Meal | Heart Prevent Meal I | Heart Prevent Meal II | Total
Number analyzed (Participants) | 42 | 41 | 39 | 122
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 24 | 16 | 23 | 63
  >=65 years | 18 | 25 | 16 | 59
Age Continuous [Mean (Standard Deviation); unit: years] | 62 (7) | 65 (8) | 62 (11) | 63 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 15 | 15 | 41
  Male | 31 | 26 | 24 | 81
Region of Enrollment [Number; unit: participants]
  Brazil | 42 | 41 | 39 | 122

OUTCOME MEASURES:

1. Primary Outcome: Systolic Blood Pressure
Description: Change From Baseline in systolic blood pressure
Time Frame: 12 weeks
Population: Participants who were evaluable at this time point were analyzed
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Brazilian Heart-prevent Meal | Heart Prevent Meal I | Heart Prevent Meal II
Number analyzed (Participants) | 40 | 41 | 39
mmHg
  Baseline | 127 (12) [-18.5 to 5.2] | 129 (16) [-6.5 to 3] | 128 (13) [-11.9 to 1.8]
  12 weeks | 117 (19) [-17.5 to -3.4] | 126 (21) [-10.1 to 1.8] | 123 (20) [-8.9 to -0.2]
Statistical Analysis 1: Comparison: Brazilian Heart-prevent Meal vs Heart Prevent Meal I vs Heart Prevent Meal II; The absolute changes has been assessed by ANOVA, in which the homogeneity of variance was assessed and the Brown-Forsythe correction was used when necessary. In cases of statistically significant differences between groups, we used multiple comparisons with Bonferroni adjustment to locate the differences. Was considered statistically significant p values <0.05. All analyzes were performed following the principle of "intention to treat."; Test type: Superiority or Other; p < 0.05, ANOVA; Mean Difference (Final Values) = 120, 95% CI [100 to 140], Standard Deviation 19

2. Secondary Outcome: Weight
Description: Change From Baseline in weight
Time Frame: 12 weeks
Population: Participants who were evaluable at this time point were analyzed
Measure: Mean (Standard Error); unit: kg
Arm/Group | Brazilian Heart-prevent Meal | Heart Prevent Meal I | Heart Prevent Meal II
Number analyzed (Participants) | 40 | 39 | 38
kg
  Baseline | 82.2 (14.9) [-3 to -1.5] | 87.9 (15.9) [-2.8 to -1] | 84.3 (15.9) [-1.5 to -0.3]
  12 weeks | 79.3 (14.9) [-4.1 to -1.7] | 85.8 (14.5) [-2.7 to -0.5] | 84.0 (16.1) [-4 to -1.7]
Statistical Analysis 1: Comparison: Brazilian Heart-prevent Meal vs Heart Prevent Meal I vs Heart Prevent Meal II; Test type: Superiority or Other; p = 0.05, ANOVA; Mean Difference (Final Values) = 78, 95% CI [66 to 95], Standard Deviation 15

3. Primary Outcome: Total Cholesterol
Description: Change From Baseline in total Cholesterol
Time Frame: 12 weeks
Population: Participants who were evaluable at this time point were analyzed.
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Brazilian Heart-prevent Meal | Heart Prevent Meal I | Heart Prevent Meal II
Number analyzed (Participants) | 40 | 41 | 39
mg/dl
  Baseline | 179 (40) | 169 (39) | 167 (35)
  12 weeks | 163 (39) | 154 (41) | 148 (30)
Statistical Analysis 1: Comparison: Brazilian Heart-prevent Meal vs Heart Prevent Meal I vs Heart Prevent Meal II; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.05, ANOVA; Mean Difference (Final Values) = 170, 95% CI [140 to 220], Standard Deviation 39

4. Secondary Outcome: Waist Circumference
Description: Change From Baseline in wais circumference
Time Frame: 12 weeks
Population: Participants who were evaluable at this time point were analyzed
Measure: Mean (Standard Error); unit: cm
Arm/Group | Brazilian Heart-prevent Meal | Heart Prevent Meal I | Heart Prevent Meal II
Number analyzed (Participants) | 40 | 41 | 39
cm
  Baseline | 102 (12) | 108 (12) | 106 (11)
  12 weeks | 99 (12) | 105 (9) | 102 (12)
Statistical Analysis 1: Comparison: Brazilian Heart-prevent Meal vs Heart Prevent Meal I vs Heart Prevent Meal II; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.05, ANOVA; Mean Difference (Final Values) = 100, 95% CI [88 to 112], Standard Deviation 12

5. Secondary Outcome: Blood Glucose
Description: Change From Baseline in blood glucose
Time Frame: 12 weeks
Population: Participants who were evaluable at this time point were analyzed
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Brazilian Heart-prevent Meal | Heart Prevent Meal I | Heart Prevent Meal II
Number analyzed (Participants) | 40 | 41 | 39
mg/dl
  Baseline | 112 (43) | 104 (22) | 108 (30)
  12 weeks | 107 (30) | 102 (20) | 112 (26)
Statistical Analysis 1: Comparison: Brazilian Heart-prevent Meal vs Heart Prevent Meal I vs Heart Prevent Meal II; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.05, ANOVA; Mean Difference (Final Values) = 100, 95% CI [77 to 137], Standard Deviation 30

ADVERSE EVENTS:
Arm/Group | Brazilian Heart-prevent Meal | Heart Prevent Meal I | Heart Prevent Meal II
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/39 | 0/38
Other Adverse Events (participants affected / at risk) | 0/40 | 0/39 | 0/38

LIMITATIONS AND CAVEATS:
Small numbers of subjects analyzed, We did not evaluate the patient's adherence to food intake, The high purchasing power of patients, Randomization with opaque envelope technique, Low statistical power.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes